CLINICAL TRIAL: NCT06290245
Title: Effect of PEP Buddy During Aerobic Training on Breathing, Exercise, and Sleep Quality in COPD Patients
Brief Title: PEP Buddy Impact on Breathing, Exercise, and Sleep Quality in COPD Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ebtesam Nabil, lecturer at Physical Therapy Department for Cardiovascular/Respiratory Disorder and Geriartics, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: P.T.REC/012/005045
Record Dates: First submitted 2024-02-21; First posted 2024-03-04 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: chronic obstructive pulmonary disease; quality of life; sleep quality; positive expiratory pressure; exercise; dyspnea
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Sleep Initiation and Maintenance Disorders; Motor Activity; Dyspnea | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- study group (Experimental): the participants will receive combined PEP Buddy plus the same exercise protocol as in the control group three times per week for eight weeks
  Interventions: Device: PEP Buddy; Other: aerobic exercise
- control group (Active Comparator): the participants will perform an aerobic exercise in the form of cycling three times per week for eight weeks
  Interventions: Other: aerobic exercise

INTERVENTIONS:
Device: PEP Buddy — It is a hands-free, oral PEP device (PEP buddy) which held by the patient's lips like a whistle and is attached to a necklace/lanyard. Different grades of PEP-buddy generate expiratory pressures of 5-17cm H2O
  Arms: study group
Other: aerobic exercise — Exercise training will start and finish with a 5-minute warm-up and cool-down on the cycle ergometers at (40% of PHR). The cycling active phase will last for 30 min. at 70% of HRmax (moderate-intensity continuous exercise).

SUMMARY:
Exercise intolerance and sleeping problems are among the most common symptoms experienced by patients with chronic obstructive pulmonary disease (COPD), which is associated with lung dynamic hyperinflation (DH). There was evidence that positive expiratory pressure (PEP), which less costly devices could offer, could reduce DH.

A positive expiratory pressure device improved COPD-related symptoms in more than 70% of patients with COPD.

PEP buddy is an adjunct to current COPD therapies, such as inhalers and pulmonary rehabilitation. It provides a tool for self-management and breathing re-training, reducing dyspnea and improving quality of life.

DETAILED DESCRIPTION:
PEP devices have been wildly used to reduce breathing frequency and expiratory flow limitation, change breathing patterns, improve gas exchange, as well as result in less airway collapse and air-trapping in patients with COPD.

Increasing COPD disease severity promotes a negative impact on exercise tolerance and magnifies the level of disability. Physical activity programs appear to safely ameliorate these COPD consequences, conferring beneficial effects on dyspnea and health-related quality of life.

The combination of PEP during aerobic exercise helps to get the most benefits from the exercise for a longer time and little dyspnea and fatigue.

ELIGIBILITY:
Inclusion Criteria:

* • All gender COPD patients

  * Age will be 55-65 years.
  * Moderate to severe COPD patients
  * emphysema on CT scan (HU ≥ - 900)
  * Their FEV1 will be less than 80% predicted
  * Class II obesity (BMI of 35 to < 40)
  * Medically stable
  * greater than 10 pack-year smoking history

Exclusion Criteria:

* • Very severe COPD - Lung cancer

  * Lung resection - Lung fibrosis
  * Heart failure - Cognitive disorders that affect the device application
  * Musculoskeletal or neurological disorders that interfere with an exercise program
  * requiring invasive or non-invasive positive pressure ventilation
  * inability to speak in complete sentences due to breathlessness
  * suspected elevated intracranial pressure - hemodynamic instability
  * recent facial, oral, or skull surgery
  * active hemoptysis (more than two tablespoons of frank blood per day)
  * pneumothorax - failure to comply with the research protocol.
  * uncontrolled hypertension, or other concomitant respiratory diseases
  * participate in any research or pulmonary rehabilitation program during the period of this study.
  * imaging changes of lung disease such as occupancy, exudation, and interstitial changes on CT scan

Ages: 55 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2024-03-23 (Actual); Primary Completion 2025-05-25 (Actual); Study Completion 2025-08-01 (Actual)

PRIMARY OUTCOMES:
dyspnea | baseline and after 8 weeks
  it will be evaluated by mMRC dyspnea scale. it is a self-rating tool to measure the degree of disability that breathlessness poses on day-to-day activities on a scale from 0 to 4: 0, no breathlessness except on strenuous exercise; 1, shortness of breath when hurrying on the level or walking up a slight hill; 2, walks slower than people of same age on the level because of breathlessness or has to stop to catch breath when walking at their own pace on the level; 3, stops for breath after walking ∼100 m or after few minutes on the level; and 4, too breathless to leave the house, or breathless when dressing or undressing

SECONDARY OUTCOMES:
pulmonary function | baseline and after 8 weeks
  by using spirometer, forced expiratory volume in the first second (FEV1), forced vital capacity (FVC), the ratio of forced expiratory volume in the first second and forced vital capacity (FEV1/FVC) will be measured
exercise capacity | baseline and after 8 weeks
  six-minute walk test is a sub-maximal exercise test that will be used to assess aerobic capacity. The distance covered over a time of 6 minutes is used as the outcome by which to compare changes in performance capacity
Sleep quality | baseline and after 8 weeks
  Sleep Quality NRS is a single-item measure that instructs the patient to "select the number that best describes the quality of his sleep during the past 24 hours," where 0 is best possible sleep and 10 is worst possible sleep
Health-related quality of life (HRQoL) | baseline and after 8 weeks
  St. George Respiratory Questionnaire is Disease-specific instrument designed to measure impact on overall health, daily life, and perceived well-being in patients with obstructive airways disease. it includes 50 items of 3 components (Part 1 : Symptoms component (frequency & severity) with a 1, 3 or 12-month recall (best performance with 3- and 12-month recall); Part 2: Activities that cause or are limited by breathlessness; Impact components (social functioning, psychological disturbances resulting from airways disease) refer to current state as the recall). Scores range from 0 to 100, with higher scores indicating more limitations.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Physical Therapy, Giza, Dokki, Egypt

IPD SHARING:
Plan to Share IPD: Undecided